CLINICAL TRIAL: NCT06430359
Title: Circadian Variation of Urinary Copper Excretion in Wilson Disease Patients Treated With Chelators or Zinc Salts
Brief Title: Circadian Variation of Urinary Copper Excretion in Wilson Disease Patients
Acronym: VARCUWIC
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_1227
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Wilson Disease
Keywords: Wilson disease; urinary copper; chelator
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Urination; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3 urine collections of an 8h period. One blood sample for liver function test and copper assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 - DP: Patients with a confirmed diagnosis of Wilson's Disease (Leipzig score ˃4 ). Aged between 6 years and 70 years. Treated with D-Pencillamine
  Interventions: Diagnostic Test: urine and blood test
- Group 2 - Trientine: Patients with a confirmed diagnosis of Wilson's Disease (Leipzig score ˃4 ). Aged between 6 years and 70 years. Treated with Trientine
  Interventions: Diagnostic Test: urine and blood test
- Group 3 - ZINC: Patients with a confirmed diagnosis of Wilson's Disease (Leipzig score ˃4 ). Aged between 6 years and 70 years. Treated with Zinc.
  Interventions: Diagnostic Test: urine and blood test

INTERVENTIONS:
Diagnostic Test: urine and blood test — 3 urine collections of an 8h period. One blood sample for liver function test and copper assessment

SUMMARY:
Wilson's disease (WD) is a genetic disorder characterized by an accumulation of copper in the body, mainly in the liver and brain. Patients suffering from this disease are monitored by liver function tests, blood copper levels, and 24-hour urinary copper determinations.

Treatment is based either on chelating the copper accumulated in the body using D-penicillamine or Trientine or on limiting intestinal copper absorption with zinc salts.

Monitoring copper elimination in urine collected over 24 hours is essential for estimating a patient's copper load, adapting treatment dosage, and detecting any copper deficiency.

Nevertheless, urine collection is often complicated for patients, given the obvious constraints of collecting urine over 24 hours. Without this, clinical decisions are usually made based on spot urine.

There is no official recommendation for monitoring urinary copper elimination other than on 24-hour urine.

According to studies on healthy volunteers under physiological conditions, urinary copper elimination occurs according to a circadian rhythm, with minimal copper elimination between 8 pm and 4 am and maximum between 8 am and noon.

The study would aim to find the period of the day best correlated with 24h urinary copper excretion

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of Wilson's Disease (Leipzig score ˃4).
* Age ≥ 6 years and ≤70 years.
* Patient able to perform 24h urine.
* Current treatment with D-Pencillamine, Trientine or Zinc.
* Non-opposition of patient and/or legal representatives for minor patients.

Exclusion Criteria:

* Patients who had a change in treatment within the last 6 months before the inclusion
* Patients who have undergone liver transplantation
* Patients with known chronic renal failure (GFR < 30 ml/min)
* Patients on long-term diuretic or corticosteroid therapy
* Persons deprived of liberty by a judicial or administrative decision
* Patient under judicial protection, unable to express consent

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Patients with a confirmed diagnosis of Wilson's Disease (Leipzig score ˃4).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-02-10 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Correlation factor | Two 24-hour urine recollection
  Correlation between 24-hour urinary copper excretion and 8-hour urinary copper excretion collected between midnight and 8 am).

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gastroentérologie, Hépatologie et Nutrition Pédiatriques - Hôpital Femme Mère Enfant, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No